CLINICAL TRIAL: NCT00445926
Title: Deep TMS With the H Coils as a Novel Strategy for the Treatment of Negative Symptoms of Schizophrenia
Brief Title: Evaluation of the H1-coil Deep TMS in the Treatment of Negative Symptoms and Cognitive Deficit in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Hilik Levkovitz, shalvataMHC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH-40206
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: deep TMS H-coil

SUMMARY:
The study evaluates the feasibility of using a 4 week stimulation protocol with the deep TMS H-coils for the treatment of negative symptoms and cognitive deficit in schizophrenia patients

ELIGIBILITY:
Inclusion Criteria:

* DSM IV Diagnosis of Schizophrenia
* PANNS Negative > 21

Exclusion Criteria:

* risk factors for convulsions
* PANNS positive > 24

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiran V Harel, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel